CLINICAL TRIAL: NCT04678037
Title: Home-based Assessment of Patient Reported Outcome (PROs) Measures in Sickle Cell Disease (SCD) Using A Smartphone App Platform: A Feasibility Study
Brief Title: Home-based Assessment of PRO Measures in SCD Using A Smartphone App Platform: A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Sherif Badawy, MD, Assistant Professor, Department of Pediatrics, Division of Hematology, Oncology and Stem Cell Transplant, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB 2017-757
Record Dates: First submitted 2020-12-03; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Sickle Cell Disease; Sickle Cell Hemoglobin C; Sickle Beta Zero Thalassemia; Sickle B+ Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell; Hemoglobin SC Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (PROs assessment every 2 weeks) (Active Comparator)
  Interventions: Behavioral: PROs assessment using sickle cell disease mobile app (SCD-app)
- Group A (PROs assessment every 4 weeks) (Active Comparator)
  Interventions: Behavioral: PROs assessment using sickle cell disease mobile app (SCD-app)

INTERVENTIONS:
Behavioral: PROs assessment using sickle cell disease mobile app (SCD-app) — A smartphone app platform designed for patients with sickle cell disease. The SCD-app is programmed to send notification to patients to complete PROs assessment. The SCD-app is able to collect PROs data as patients complete the assessment using the app platform.

SUMMARY:
The overarching goal of this proposal is to identify modifiable behavioral strategies based on patient-reported outcomes (PROs) and health-related quality of life (HRQOL) that will improve hydroxyurea (HU) adherence among adolescents and young adults with sickle cell disease (SCD). In this proposed study, we intend to test the functionality of a PROs-toolbox feature, which will be integrated into our existing smartphone application platform (SCD-app), over a 24-week period in a cohort of SCD patients and their caregivers.

DETAILED DESCRIPTION:
Adherence to hydroxyurea is a multi-factorial dynamic process, and, to date, predictors for changes in adherence levels over time remain unclear. Changes in HRQOL data could serve as surrogate markers for changes in hydroxyurea adherence over time, and could suggest when patients might or might not need or benefit from an intervention based on worse or better HRQOL scores, respectively.

The main hypothesis of this study is that the assessment of patients' HRQOL at home using a SCD smartphone application platform (app) is feasible and acceptable, and that less frequent assessments of HRQOL at home will have an overall higher completion rate when compared to more frequent ones. We plan to assess HRQOL using the NIH-developed patient reported outcomes measurement information system (PROMIS®) with computerized adaptive testing (CAT) approach. PROMIS®-CAT approach is a reliable and valid PROs assessment platform that has been used in limited studies in SCD.

The study will include the following specific aims:

1. To evaluate the feasibility and acceptability of the assessment of patients HRQOL at home using smartphones with PROMIS®-CAT measures integrated into a SCD-app.
2. To examine the effect of the frequency of required HRQOL assessments on participants' completion rate over 24-week period with HRQOL evaluated every 2 weeks (Group 1) versus every 4 weeks (Group 2).
3. To explore participants' experience and preferences with the process and the frequency of HRQOL assessment at home using their smartphones with PROMIS®-CAT measures integrated into a SCD-app.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years or older at the time of study enrollment;
* SCD diagnosis (all genotypes) confirmed by hemoglobin electrophoresis;
* Own or have access to a smartphone or a tablet; and
* Speak and read English.

Exclusion Criteria:

* Patients or caregivers with cognitive impairment;
* Patients or caregivers physical impairment; and
* Patients or caregivers who will not be able to complete study assessments.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-07-21 (Actual); Study Completion 2019-07-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of completing PRO assessments at home using SCD-app (HU-Go) | 6 months
  Having an overall completion rate of ≥ 50% for all study participants (Group A and B). This will be reported as a dichotomous outcome, either yes or no. The percentage (%) completion rate will be calculated as the number of PROs assessments completed divided by the number of PROs assessments expected over the study period.

SECONDARY OUTCOMES:
Completion rate of PRO assessments at home using SCD-app (HU-Go) | 6 months
  Completion rate of different PRO assessments at home using PROMIS®-CAT measures among patients with SCD and/or their parents. PRO assessments are planned to be every 2 weeks in Group 1 and every 4 weeks in Group 2. This outcome will be calculated and reported as percent (%) completion rate.

CONTACTS AND LOCATIONS:
Overall Officials: Sherif M Badawy, MD, MS, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
All study data are de-identified and will be analysed as aggregate.